CLINICAL TRIAL: NCT06838117
Title: From Variability to Standardization: The Impact of Breast Density on Background Parenchymal Enhancement in Contrast-Enhanced Mammography and the Need for a Structured Reporting System
Status: Enrolling by invitation | Type: Observational
Sponsor: Graziella di Grezia (Other)
Collaborators: Link Campus University (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor-Investigator, Graziella di Grezia, Principal Investigator, Link Campus University
Organization: Link Campus University (Other)
Other Study IDs: T_5_2025
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: To Establish a Standardized Background Parenchimal Enhancement Classification System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Cohort of Women Undergoing Contrast-Enhanced Mammography (CEM) for Diagnostic and Surv

SUMMARY:
This retrospective study includes 213 patients who underwent CEM, mammography (MG), and ultrasound (US) between May 2022 and June 2023 at the P.O. 'A. Perrino' Hospital, Brindisi. BPE was categorized into four levels (Minimal, Light, Moderate, and Marked), while breast density was rated according to the ACR BI-RADS (A-D) classification. A statistical analysis was performed to assess the correlation between BPE and breast density, supporting the development of the BPE-CEM Standard Scale (BCSS) to standardize reporting and improve interobserver agreement.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent CEM, mammography, and ultrasound between May 2022 and June 2023.

Availability of BPE assessment and BI-RADS density classification.

Complete imaging dataset available for analysis.

Exclusion Criteria:

Patients with prior breast cancer treatment that could alter BPE.

Incomplete imaging data or missing classification values.

Contraindications to contrast-enhanced imaging.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years and older who underwent CEM for diagnostic or surveillance purposes.
  Patients with recorded BPE levels and BI-RADS breast density classification.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between breast density and background parenchymal enhancement (BPE) in CEM. | Data analysis within 12 months of study completion.
  This outcome assesses whether increased breast density is associated with higher BPE levels and evaluates the statistical significance of the correlation.

SECONDARY OUTCOMES:
Development and validation of the BPE-CEM Standard Scale (BCSS). | Within 12 months of study completion.
  Establishing a structured lexicon for BPE classification and assessing its clinical utility.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Di Grezia, Medicine and Surgery, Principal Investigator — Link Campus University
Locations (1):
- Pellino Hospital, Brindisi, Italy

IPD SHARING:
Plan to Share IPD: No